CLINICAL TRIAL: NCT02196324
Title: A Randomized, Double-Blind, Placebo-Controlled, Study of Neurokinin-1 Receptor Antagonist Serlopitant in Subjects With Prurigo Nodularis
Brief Title: A Randomized Placebo-Controlled Study of the Neurokinin-1 (NK1) Receptor Antagonist Serlopitant Prurigo Nodularis (PN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCP-102
Record Dates: First submitted 2014-07-14; First posted 2014-07-22 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo Nodularis; Atopic Dermatitis; Lichen-simplex chronicus
MeSH Terms: conditions — Dermatitis, Atopic; Lichenoid Eruptions | interventions — serlopitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- serlopitant 5 mg tablets (Active Comparator): serlopitant 5 mg tablets
  Interventions: Drug: serlopitant
- Placebo tablets (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: serlopitant — NK1 receptor antagonist
  Other Names: VPD-737
  Arms: serlopitant 5 mg tablets
Drug: Placebo — Placebo
  Arms: Placebo tablets

SUMMARY:
The purpose of this study is to demonstrate whether or not VPD-737, an NK1 receptor antagonist is safe and effective for treatment of prurigo nodularis versus placebo.

DETAILED DESCRIPTION:
The sensation of itch is transmitted to the brain through the nervous system. Several chemicals are involved in transmitting this signal.This trial of VPD 737 is intended to treat this condition by blocking one of the chemicals involved in the transmission of the itch signal. This is an oral drug administered once daily It has been used in other trials and has shown to be safe at the doses used in this trial. The trial will involve once daily pills for 8 weeks. Subject will be asked to fill out questionnaires both electronically and on paper during the study period. Patients will also be monitored for safety and will have blood taken for testing and several points during the trial. Overall participation will last about 14 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria will be eligible for study entry:

  1. Males or females who are at least 18 years and no more than 80 years of age at Screening.
  2. Must have PN (defined as the presence of pruritic nodules due to chronic pruritus,) of more than 6 weeks duration despite treatment with current therapies such as antihistamines or corticosteroids ("treatment resistant" PN).
  3. Must have PN lesions on both arms, both legs, and/or the trunk (ie, the lesions must not be localized).
  4. Must have a VAS pruritus score of 70 or greater within 72 hours of Baseline.
  5. Males, non-fecund females (ie, surgically sterilized, if procedure was done 12 months before screening or subject is postmenopausal, without menses for 12 months before screening), or females of childbearing potential using an acceptable method of birth control for a period of 35 days before the first dosing, and all females must have a negative pregnancy test at the screening and baseline visits:

     Note 1: Acceptable methods of birth control include any one of the following:

     abstinence, vasectomized sexual partner, hormonal methods (ie, birth-control pill, hormonal IUD, Depo-Provera, implants, patch, intravaginal device [NuvaRing]), intrauterine device (IUD [copper banded coils]), diaphragm, cervical cap, or condom with spermicidal jelly or foam. Subjects using oral contraceptives must also use a reliable backup method of birth control during the study and until the first menses after the last dose of study medication or for 14 days menses after the last dose of study medication.
  6. Willing and able to understand and provide written informed consent.
  7. Willing and able to comply with study requirements and restrictions including the discontinuation of all current therapies for pruritus.
  8. Subjects must be in good health as determined by medical history, physical examination, and results of Electro Cardio Gram (ECG) and clinical laboratory tests (including urinalysis).
  9. Agreeing to confidential use and storage of all data and use of all anonymized data for publication including scientific publication.

Exclusion Criteria:

* Subjects not eligible for the study are those who:
* Have chronic pruritus due conditions other than PN, such as the following conditions:
* Lichen simplex chronicus
* Lichen amyloidosus
* Localized pruritus (e.g., only one arm affected)
* Neuropathic and psychogenic pruritus (notalgia paresthetica, brachioradial pruritus, somatoform prurigo, dilusional parasitosis, depression associated prurigo)
* Active dermatoses needing immediate therapy such as atopic dermatitis (without PN) or bullous pemphigoid;
* Have a history of use (within the specified time periods) of the medications listed below. Prior to randomization, a subject who used any of these medications must undergo a washout period equal to the length of the interval specified below (eg, 2 weeks for antihistamines, 4 weeks for naltrexone, and 4 weeks for cyclosporine A).
* Topical or systemic antihistamines, (used ≤2 weeks prior to the baseline visit) [loratindine, or cetirizine may act as rescue medication during treatment];
* Topical calcineurin inhibitors, topical capsaicin, menthol, camphor, polidocanol, topical antibiotics, antiseptic baths and cleansing lotions (used ≤2 weeks prior to the baseline visit);
* Topical steroids (used ≤2 weeks prior to the baseline visit);
* Naltrexone, paroxetine, fluvoxamine, amitriptyline, gabapentin, pregabalin, or UVtherapy (prescribed for the pruritus treatment) (used ≤4 weeks prior to the baseline visit);
* Systemic steroids (used ≤4 weeks prior to the baseline visit);
* Cyclosporine A and other immunosuppressants (used ≤4 weeks prior to the baseline visit).
* Have any medical condition or disability that would interfere with the assessment of safety or efficacy in this trial or would compromise the ability of the subject to undergo study procedures or to give informed consent.
* Have any chronic or acute medical condition that, in the opinion of the investigator, might interfere with the study results or place the subject at undue risk.
* Have a history of sensitivity to any components of the study material.
* Are females of childbearing potential who are unwilling to use adequate contraception or who are breast feeding.
* Have chronic renal disease, ie, serum creatinine greater than 2.4 mg/dL.
* Have aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2 times the upper limit of normal. Subjects with hepatitis B or C who have normal liver function may be enrolled.
* Have a current malignancy (such as Hodgkin's lymphoma, B or T cell lymphoma, or myeloma) or blood cell dyscrasia (eg, polycythemia or myelofibrosis) that might lead to systemic chronic pruritus.
* Subjects with untreated hyperthyroidism.
* Have pruritus of psychiatric etiology (eg, delusions of parasitosis, obsessive compulsive disorder, or major depression) or neuropathic etiology (eg, due to shingles, spinal cord injury or with neurologic deficit).
* Have pruritus due to urticaria, drug allergy, or infection (such as pityriasis rosea or tinea or active human immunodeficiency virus [HIV]). Note: Subjects with HIV who have undetectable viral load, CD 4 counts >200 cells/cc, and stable retroviral therapy may enroll.
* Are on medications known to cause pruritus (ie, Erbitux®, opioids, cocaine, amphetamines, and angiotensin converting enzyme [ACE] inhibitors) and are suspected of having drug-induced pruritus.
* Have taken investigational medications within 30 days prior to Screening.
* Are currently participating in any other clinical study.
* Have a history (within the previous 4 weeks) of use of tricyclic antidepressants, selective serotonin reuptake inhibitors (SSRI), serotonin-norepinephrine reuptake inhibitors (SNRIS), monoamine oxidase (MAO) inhibitors, opioids, immunemodulators (e.g. azathioprine, methotrexate, mycophenolate mofetil, cyclosporine A, antibodies), or neuroactive medications (e.g. pregabalin, gabapentin).
* Have a history (within the previous 4 weeks) of use of sedatives or tranquilizers.

Subjects must undergo an appropriate washout period from any sedatives or tranquilizers before enrolling in the study.

* Are currently treated with strong CYP3A4 inhibitors (e.g. conazole, ketoconazole, fluconazole, itraconazole, voroconazole etc. or erythromycin). The co-administration of moderate CYP3A4 inhibitors to VPD-737 may be allowed with investigator agreement and appropriate safety monitoring.
* Received ultraviolet B (UVB) or psoralen + ultraviolet A (PUVA) treatment within 30 days prior to Screening.
* Within the past 12 months, have expressed suicidal ideation with some intent to act.
* Started or changed creams, or emollients including over-the-counter (OTC) preparations or bath oil treatment for relief of pruritus within 2 weeks prior to Screening.
* Have any social or medical condition (eg, alcoholism, drug dependency, psychotic state) that, in the investigator's opinion, might interfere with the subject's ability to comply with the requirements of the protocol.
* Are employees of the study site or of the Sponsor's company.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Staender, MD, Principal Investigator — University of Muenster, Germany
Locations (15):
- Germany (15):
  - Study Site 08, Bonn
  - Study Site 06, Dresden
  - Study Site 12, Düsseldorf
  - Study Site 02, Frankfurt
  - Study Site 09, Hamburg
  - Study Site 05, Heidelberg
  - Study Site 03, Kiel
  - Study Site 11, Leipzig
  - Study Site 04, Lübeck
  - Study Site 14, Mainz
  - Study Site 07, Mitte
  - Study Site 16, München
  - Study Site 01, Münster
  - Study Site 15, Selters
  - Study Site 10, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimel M, Zeidler C, Kwon P, Revicki D, Stander S. Validation of Psychometric Properties of the Itch Numeric Rating Scale for Pruritus Associated With Prurigo Nodularis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2020 Dec 1;156(12):1354-1358. doi: 10.1001/jamadermatol.2020.3071. PMID 32936233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were randomized at 15 sites in Germany.
Pre-assignment Details: This study consisted of a screening period of up to 4 weeks. All the assessments were done at screening as per the schedule of assessment.
Groups:
- Placebo: Randomized participants took matching placebo tablets for oral administration as 3 tablets at baseline (Day 1) followed by 1 tablet every day at bedtime for 8 weeks.
- Serlopitant: Randomized participants took Serlopitant 5 mg tablets for oral administration at a loading dose of 3 tablets at baseline (Day 1) followed by 1 tablet every day at bedtime for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Serlopitant
Started | 63 | 65
Completed | 48 | 57
Not Completed | 15 | 8
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Adverse Event or Serious Adverse Event | 6 | 3
Not completed — Occurrence of an Exclusion Criterion | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population - all randomized participants who were treated. This population was analyzed based upon the treatment to which participants were randomized.
  Of the 128 randomized participants, 127 received study drug (63 placebo, 64 serlopitant) and comprised the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Serlopitant | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (11.14) | 57.1 (12.00) | 57.6 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 31 | 67
  Male | 27 | 33 | 60

OUTCOME MEASURES:

1. Primary Outcome: Average Visual Analog Scale at Baseline
Description: At study visits, participants recorded a mark for pruritus severity on a 10-cm horizontal line. This thermometer-type scale was marked with ratings of "no itch" (0 cm) and worst imaginable itch" (10 cm). Average Visual Analog Scale (VAS) (average itch over the past 24 hours) was recorded. Higher scores indicated worse outcome.
Time Frame: At Baseline
Population: The Intent-to-treat (ITT) population - all randomized participants who were treated. This population was analyzed based upon the treatment to which participants were randomized.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Units on a scale | 7.92 (1.630) | 7.88 (1.311)

2. Primary Outcome: Average Visual Analog Scale at Week 2
Description: At study visits, participants recorded a mark for pruritus severity on a 10-cm horizontal line. This thermometer-type scale was marked with ratings of "no itch" (0 cm) and worst imaginable itch" (10 cm). Average VAS (average itch over the past 24 hours) was recorded. Higher scores indicated worse outcome.
Time Frame: At Week 2
Population: The ITT population - all randomized participants who were treated. This population was analyzed based upon the treatment to which participants were randomized.
  Here, overall number of participants analyzed signifies only the participants with available data that were analyzed for the outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 61 | 63
Units on a scale | 7.01 (2.187) | 6.06 (2.236)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant; Test type: Superiority; p = 0.0111, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.5 to -0.2], Standard Error of Mean 0.34

3. Primary Outcome: Average Visual Analog Scale at Week 4
Description: as for outcome 2
Time Frame: At Week 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 54 | 64
Units on a scale | 6.32 (2.403) | 5.41 (2.719)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant; Test type: Superiority; p = 0.0248, Mixed Models Analysis; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.8 to -0.1], Standard Error of Mean 0.43

4. Primary Outcome: Average Visual Analog Scale at Week 8
Description: as for outcome 2
Time Frame: At Week 8
Population: Intent-to-treat (ITT) population - all randomized participants who were treated. This population was analyzed based upon the treatment to which participants were randomized.
  Here, overall number of participants analyzed signifies only the participants with available data that were analyzed for the outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 46 | 57
Units on a scale | 5.56 (2.630) | 4.21 (2.746)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.6 to -0.7], Standard Error of Mean 0.47

5. Secondary Outcome: Number of Participants With Improvement in Pruritus as Reported on Verbal Rating Scale (VRS) - Pruritus
Description: At study visits, participants used the VRS to rate their skin sensations (pruritus, burning, and stinging) using a 5-point scale (0 = not present; 1 = mild present; 2 = moderately present; 3 = severely present; and 4 = very severely present). Higher scores indicated worse outcome.
Time Frame: At Baseline and Week 8
Population: The ITT population - all randomized participants who were treated. This population was analyzed based upon the treatment to which participants were randomized.
  Here, number analyzed in each row signifies only the participants with available data that were analyzed for each parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Participants
  Baseline, Mild Present: number analyzed (Participants) | 62 | 64
  Baseline, Mild Present | 2 | 0
  Baseline, Moderately Present: number analyzed (Participants) | 62 | 64
  Baseline, Moderately Present | 18 | 17
  Baseline, Severely Present: number analyzed (Participants) | 62 | 64
  Baseline, Severely Present | 20 | 32
  Baseline, Very Severely Present: number analyzed (Participants) | 62 | 64
  Baseline, Very Severely Present | 22 | 15
  Week 8, Not Present: number analyzed (Participants) | 45 | 57
  Week 8, Not Present | 2 | 4
  Week 8, Mild Present: number analyzed (Participants) | 45 | 57
  Week 8, Mild Present | 11 | 27
  Week 8, Moderately Present: number analyzed (Participants) | 45 | 57
  Week 8, Moderately Present | 18 | 17
  Week 8, Severely Present: number analyzed (Participants) | 45 | 57
  Week 8, Severely Present | 9 | 7
  Week 8, Very Severely Present: number analyzed (Participants) | 45 | 57
  Week 8, Very Severely Present | 5 | 2

6. Secondary Outcome: Number of Participants With Improvement in Burning as Reported on Verbal Rating Scale (VRS) - Burning
Description: as for outcome 5
Time Frame: At Baseline and Week 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Participants
  Baseline, Not Present: number analyzed (Participants) | 62 | 64
  Baseline, Not Present | 14 | 21
  Baseline, Mild Present: number analyzed (Participants) | 62 | 64
  Baseline, Mild Present | 8 | 5
  Baseline, Moderately Present: number analyzed (Participants) | 62 | 64
  Baseline, Moderately Present | 13 | 21
  Baseline, Severely Present: number analyzed (Participants) | 62 | 64
  Baseline, Severely Present | 18 | 12
  Baseline, Very Severely Present: number analyzed (Participants) | 62 | 64
  Baseline, Very Severely Present | 9 | 5
  Week 8, Not Present: number analyzed (Participants) | 43 | 56
  Week 8, Not Present | 11 | 31
  Week 8, Mild Present: number analyzed (Participants) | 43 | 56
  Week 8, Mild Present | 9 | 10
  Week 8, Moderately Present: number analyzed (Participants) | 43 | 56
  Week 8, Moderately Present | 15 | 8
  Week 8, Severely Present: number analyzed (Participants) | 43 | 56
  Week 8, Severely Present | 5 | 6
  Week 8, Very Severely Present: number analyzed (Participants) | 43 | 56
  Week 8, Very Severely Present | 3 | 1

7. Secondary Outcome: Number of Participants With Improvement in Stinging as Reported on Verbal Rating Scale (VRS) - Stinging
Description: as for outcome 5
Time Frame: At Baseline and Week 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Participants
  Baseline, Not Present: number analyzed (Participants) | 62 | 64
  Baseline, Not Present | 26 | 21
  Baseline, Mild Present: number analyzed (Participants) | 62 | 64
  Baseline, Mild Present | 8 | 14
  Baseline, Moderately Present: number analyzed (Participants) | 62 | 64
  Baseline, Moderately Present | 11 | 16
  Baseline, Severely Present: number analyzed (Participants) | 62 | 64
  Baseline, Severely Present | 9 | 10
  Baseline, Very Severely Present: number analyzed (Participants) | 62 | 64
  Baseline, Very Severely Present | 8 | 3
  Week 8, Not Present: number analyzed (Participants) | 43 | 54
  Week 8, Not Present | 18 | 30
  Week 8, Mild Present: number analyzed (Participants) | 43 | 54
  Week 8, Mild Present | 8 | 12
  Week 8, Moderately Present: number analyzed (Participants) | 43 | 54
  Week 8, Moderately Present | 10 | 7
  Week 8, Severely Present: number analyzed (Participants) | 43 | 54
  Week 8, Severely Present | 4 | 4
  Week 8, Very Severely Present: number analyzed (Participants) | 43 | 54
  Week 8, Very Severely Present | 3 | 1

8. Secondary Outcome: Worst Visual Analog Scale (VAS)
Description: At study visits, participants recorded a mark for pruritus severity on a 10-cm horizontal line. This thermometer-type scale was marked with ratings of "no itch" (0 cm) and worst imaginable itch" (10 cm). Worst VAS (worst itch over the past 24 hours) was recorded. Higher scores indicated worse outcome.
Time Frame: At Baseline, Weeks 2, 4, and 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Units on a scale
  Baseline | 8.75 (1.316) | 8.43 (1.190)
  Week 2: number analyzed (Participants) | 61 | 63
  Week 2 | 7.92 (1.733) | 6.85 (2.157)
  Week 4: number analyzed (Participants) | 54 | 64
  Week 4 | 7.46 (2.285) | 6.19 (2.690)
  Week 8: number analyzed (Participants) | 46 | 57
  Week 8 | 6.73 (2.591) | 4.82 (2.729)

9. Secondary Outcome: Number of Participants With Improvement in Pruritus as Reported on Patient Global Assessment (PGA)
Description: The PGA included a question: Did the pruritus improve during the treatment period (yes/no).
Time Frame: At Weeks 2, 4, and 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Participants
  Week 2: number analyzed (Participants) | 61 | 63
  Week 2 | 23 | 37
  Week 4: number analyzed (Participants) | 54 | 64
  Week 4 | 29 | 43
  Week 8: number analyzed (Participants) | 46 | 57
  Week 8 | 25 | 47

10. Secondary Outcome: Numeric Rating Scale (NRS)
Description: Numeric Rating Scale: Using the patient diary, participants rated the following using an 11-point NRS (0 = no itching; to 10 = worst itch imaginable): average itching over the past 24 hours (Average NRS). Higher scores indicated worse outcome.
Time Frame: At Baseline, Weeks 2, 4, and 8
Population: The ITT population - all randomized participants who were treated. This population was analyzed based upon the treatment to which participants were randomized.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Units on a scale
  Baseline: number analyzed (Participants) | 48 | 48
  Baseline | 7.65 (1.669) | 7.60 (1.455)
  Week 2: number analyzed (Participants) | 58 | 62
  Week 2 | 6.23 (2.043) | 5.50 (1.944)
  Week 4: number analyzed (Participants) | 52 | 62
  Week 4 | 5.80 (2.133) | 4.91 (2.158)
  Week 8: number analyzed (Participants) | 46 | 54
  Week 8 | 5.11 (2.320) | 4.02 (2.190)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant; Week 2; Test type: Superiority; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.4 to -0.0]
Statistical Analysis 2: Comparison: Placebo vs Serlopitant; Week 4; Test type: Superiority; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.7 to -0.1]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant; Week 8; Test type: Superiority; p = 0.0175, t-test, 2 sided — p-value assume equal variance; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.0 to -0.2]

11. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: At each visit, participants completed a DLQI questionnaire. The DLQI is a validated questionnaire consisting of 10 questions relating to the degree to which the participant's skin condition affected his/her daily activities. The DLQI questionnaire is designed for use in adults, i.e. participants over the age of 16.
  The scoring of each question is as follows:
  Very much: scored 3, A lot: scored 2, A little: scored 1, Not at all: scored 0, Not relevant: scored 0, Question 7, 'prevented work or studying': scored 3.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  Interpreting the DLQI Scores:
  0 - 1: no effect at all on participant's life, 2 - 5: small effect on participant's life, 6 - 10: moderate effect on participant's life, 11 - 20: very large effect on participant's life, 21 - 30: extremely large effect on participant's life.
Time Frame: At Baseline, Weeks 2, 4, and 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Units on a scale
  Baseline: number analyzed (Participants) | 61 | 61
  Baseline | 14.9 (7.03) | 13.7 (6.76)
  Week 2: number analyzed (Participants) | 57 | 62
  Week 2 | 12.4 (6.94) | 11.6 (6.20)
  Week 4: number analyzed (Participants) | 51 | 62
  Week 4 | 11.6 (6.56) | 11.4 (6.80)
  Week 8: number analyzed (Participants) | 44 | 55
  Week 8 | 11.3 (6.83) | 10.6 (7.31)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant; Week 2; Test type: Superiority; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.1 to 1.6]
Statistical Analysis 2: Comparison: Placebo vs Serlopitant; Week 4; Test type: Superiority; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.7 to 2.3]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant; Week 8; Test type: Superiority; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-3.6 to 2.1]

12. Secondary Outcome: Pruritus-specific Quality of Life (ItchyQoL)
Description: At each visit, participants completed an ItchyQoL questionnaire. The ItchyQoL is a validated questionnaire consisting of 22 questions based on the concerns and issues pertinent to participants with pruritus.
  Items should be scored for the following answers:
  Never: 1, Rarely: 2, Sometimes: 3, Often: 4, All the time:5. Higher scores indicated worse outcome. Total Score is obtained by calculating the unweighted mean of all ItchyQoL questions.
Time Frame: At Baseline, Weeks 2, 4, and 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Units on a scale
  Baseline | 3.68 (0.737) | 3.52 (0.679)
  Week 2: number analyzed (Participants) | 61 | 63
  Week 2 | 3.50 (0.795) | 3.36 (0.670)
  Week 4: number analyzed (Participants) | 54 | 64
  Week 4 | 3.36 (0.863) | 3.26 (0.730)
  Week 8: number analyzed (Participants) | 46 | 57
  Week 8 | 3.33 (0.876) | 3.09 (0.904)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant; Week 2; Test type: Superiority; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs Serlopitant; Week 4; Test type: Superiority; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Serlopitant; Week 8; Test type: Superiority; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.6 to 0.1]

13. Secondary Outcome: Patient Benefit Index, Version for Patients With Pruritus (PBI-P)
Description: At Visits 2 and 5 (or Early termination) only, participants completed the standardized and validated PBI-P questionnaire. Prior to treatment, the first page of the questionnaire, the Patient Needs Questionnaire (PNQ), was administered to determine how different benefits of therapy were relevant for the individual participant. After treatment, using the Patient Benefit Questionnaire (PBQ), participants were asked to evaluate the extent to which the benefits they indicated were important to them were, in fact, realized. From all the items taken together, a weighted total benefit value was calculated, which represented the patient relevant therapy benefits. The mean score greater than 1 is considered to represent a clinically relevant improvement. The items are rated on a 5-point scale with values from 0 (not at all) to 4 (very), allowing for "does/did not apply to me" = 5; and missing value = -9. Higher scores indicated better outcome.
Time Frame: At Week 8 / End of Treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 61 | 63
Units on a scale | 0.81 (0.984) | 1.16 (1.095)
Statistical Analysis 1: Comparison: Placebo vs Serlopitant; Test type: Superiority; p = 0.0625, t-test, 2 sided — p-value assume equal variance; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.02 to 0.72]

14. Secondary Outcome: Number of Participants With Improvement in PN Lesions as Reported on Investigator Global Assessment (IGA)
Description: Using the IGA, physicians rated change in PN lesions (if any) from +5 ("markedly improved") to -5 ("markedly worse"). Higher scores indicated better outcome.
Time Frame: At Week 8
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 47 | 57
Participants
  Markedly Improved | 0 | 4
  Largely Improved | 2 | 3
  Moderately To Largely Improved | 4 | 3
  Moderately Improved | 4 | 11
  Mildly Improved | 9 | 17
  Baseline | 14 | 7
  Mildly Worse | 8 | 5
  Moderately Worse | 4 | 4
  Moderately To Largely Worse | 1 | 1
  Largely Worse | 1 | 2

15. Secondary Outcome: Number of Participants With Improvement on Prurigo Activity Score (PAS)
Description: Using the PAS, physicians described, localized, counted, and measured PN lesions.
  One of the 7 items was:
  Activity Stage (Stage 0-4: 0 = 0%, 1 = 1-25%, 2 = 26-50%, 3 = 51-75%, 4 = > 75%)
  a. Prurigo lesions with excoriations/crusts
  Participants with PAS activity stage (prurigo lesions with excoriations/crusts) is presented in the below table.
Time Frame: At Day 1 and Week 8
Population: The ITT population - all randomized participants who were treated. This population was analyzed based upon the treatment to which participants were randomized.
  Here, number analyzed in each row signifies only the participants with available data that were analyzed for each day and week.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Participants
  Day 1, 1 - 25 % | 7 | 5
  Day 1, 26 - 50 % | 18 | 19
  Day 1, 51 - 75 % | 17 | 19
  Day 1, >75 % | 21 | 21
  Week 8, 0 %: number analyzed (Participants) | 47 | 57
  Week 8, 0 % | 0 | 4
  Week 8, 1 - 25 %: number analyzed (Participants) | 47 | 57
  Week 8, 1 - 25 % | 11 | 15
  Week 8, 26 - 50 %: number analyzed (Participants) | 47 | 57
  Week 8, 26 - 50 % | 12 | 12
  Week 8, 51 - 75 %: number analyzed (Participants) | 47 | 57
  Week 8, 51 - 75 % | 11 | 11
  Week 8, >75 %: number analyzed (Participants) | 47 | 57
  Week 8, >75 % | 13 | 15

16. Secondary Outcome: Participants With Rescue Medication Usage
Description: Rescue medications included cetirizine hydrochloride, desloratadine, levocetirizine, and loratadine.
Time Frame: Pre-treatment, upto 8 Weeks
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Participants
  Pre-treatment Rescue Medication Used | 15 | 17
  Used Rescue Medication | 12 | 8

17. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE (also referred to as an adverse experience) could be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, without any judgment about causality.
Time Frame: From the time of informed consent (Screening) until the last study visit (follow-up phone call, Week 10)
Population: Safety population - participants who received at least one dose of study drug. This population was analyzed based upon the actual treatment received. Participants with dosing errors were assigned to a treatment group based upon the treatment they received most often.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Serlopitant
Number analyzed (Participants) | 63 | 64
Participants
  Participants with AEs | 39 | 46
  Participants with Treatment-emergent adverse events (TEAEs) | 39 | 46
  Participants with TEAEs leading to discontinuation | 6 | 3
  Participants with TEAEs related to study drug | 22 | 31
  Participants with TEAEs by maximum severity, Mild | 14 | 18
  Participants with TEAEs by maximum severity, Moderate | 22 | 22
  Participants with TEAEs by maximum severity, Severe | 3 | 6
  Participants with serious TEAEs | 2 | 3

ADVERSE EVENTS:
Time Frame: From the time of informed consent (Screening) until the last study visit (follow-up phone call, Week 10).
Arm/Group | Placebo | Serlopitant
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 2/63 | 3/64
Other Adverse Events (participants affected / at risk) | 20/63 | 31/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Serlopitant (N=64)
Bradycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic elastosis (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Serlopitant (N=64)
Diarrhoea (Gastrointestinal disorders) | 3 | 7
Fatigue (General disorders) | 4 | 6
Oedema peripheral (General disorders) | 0 | 4
Nasopharyngitis (Infections and infestations) | 2 | 11
Urinary tract infection (Infections and infestations) | 4 | 0
Dizziness (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days